CLINICAL TRIAL: NCT02139735
Title: Therapeutic Response of Ultrasound and Muscular Stretching in Temporomandibular Disorder Patients: Clinical Trial
Brief Title: Therapeutic Response of Ultrasound and Muscular Stretching in Temporomandibular Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Eliane Correa, Doctor, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UFSM-MO-01
Record Dates: First submitted 2014-05-09; First posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders,; Ultrasonics,; Electromyography,; Pain Measurement,; Muscle Stretching Exercise
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ultrasound (Experimental): 3 MHz (Mega Hertz) ultrasound in continuous mode with an intensity of 1.0 W / cm ² was applied for 3 minutes in the TMJ (Temporomandibular joint) and masseter muscles bilaterally
  Interventions: Other: Ultrasound associated with stretching; Other: Placebo
- Ultrasound associated with stretchting (Experimental): 3 MHz ultrasound in continuous mode with an intensity of 1.0 W / cm ² was applied for 3 minutes in the TMJ and masseter muscles bilaterally.
  Active stretching of the masseter muscles with mouth opening and closed lips
  Interventions: Other: Ultrasound; Other: Placebo
- Placebo (Experimental): Turned off ultrasound application on area of TMJ and masseter muscle, bilaterally.
  Interventions: Other: Ultrasound; Other: Ultrasound associated with stretching

INTERVENTIONS:
Other: Ultrasound — 3 MHz ultrasound in continuous mode with an intensity of 1.0 W / cm ² was applied for 3 minutes in the TMJ and masseter muscles bilaterally
  Arms: Placebo; Ultrasound associated with stretchting
Other: Ultrasound associated with stretching — 3 MHz ultrasound in continuous mode with an intensity of 1.0 W / cm ² was applied for 3 minutes in the TMJ and masseter muscles, bilaterally.
  Active stretching of the masseter muscles with mouth opening and closed lips
  Arms: Placebo; Ultrasound
Other: Placebo — Turned off ultrasound application on area of TMJ and masseter muscle, bilaterally.
  Arms: Ultrasound; Ultrasound associated with stretchting

SUMMARY:
The combination of ultrasound and muscular stretching may have positive effects on pain relief and on the balance of the masticatory muscles activity.

DETAILED DESCRIPTION:
This study aimed to evaluate the therapeutic response of ultrasound (US) and ultrasound associated with stretching of the masticatory muscles on the pressure pain threshold and the electrical activity of masseter and anterior temporal muscles in Temporomandibular Disorder (TMD) patients . The study included 18 women with TMD diagnosed by the instrument Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD). The pressure pain threshold, evaluated through algometry, and the electrical activity of the masticatory muscles were evaluated, by means of surface electromyography, before and immediately after the therapeutic procedures. The volunteers underwent three different interventions: ultrasound, ultrasound associated with stretching and ultrasound placebo, with a 1-week of minimum interval between them.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of myogenic or mixed TMD according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC / TMD)
* women aged 20 to 35 years.

Exclusion Criteria:

* psychomotor impairment ;
* history of orthopedic trauma involving the temporomandibular region , orofacial surgery or poor training ;
* analgesics , anti-inflammatories , muscle relaxants , antidepressants ;
* presence of acute TMJ pain ( last 3 months) ;
* have perform physical therapy or speech therapy for the past 6 months;
* periods of the end of the menstrual cycle (7 days prior to menstruation ) and onset of menstruation ( first 2 days ) were excluded for conducting evaluations of volunteers who did not use oral contraception and those who used it to break.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | 10 minutes
  algometry

SECONDARY OUTCOMES:
surface electromyography | 10 minutes
  electromyographic activity was measure at rest, in maximal intercuspal position and maximal voluntary clench

CONTACTS AND LOCATIONS:
Overall Officials: Eliane C. Corrêa, Doctor, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Universidade Federal de Santa Maria, Santa Maria, Rio Grande do Sul, Brazil